CLINICAL TRIAL: NCT03120858
Title: Reliability and Validity of the Turkish Version of the Kinesthetic and Visual Imagery Questionnaire
Brief Title: Turkish Version of the Kinesthetic and Visual Imagery Questionnaire
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Burcu Dilek, PT, MS, PhD, Assist Prof, Hacettepe University
Other Study IDs: GO 14/568
Record Dates: First submitted 2017-04-16; First posted 2017-04-19 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Image, Body; Healthy; Pain
Keywords: motor imagery; kinesthetic imagery; reliability; Turkish version
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Determine what the imagery levels are — Determine the motor imagery: kinesthetic and visual imagery
  Other Names: Determine the motor imagery

SUMMARY:
Imagery is determined with two strategies to mentally simulate the movements: visual and kinesthetic imagery. Visual motor imagery (VMI) is associated with spatial coordinates of a movement in the environment and through this speciality VMI applies mainly to the imagery of moving objects or to movement of another person in the imagined environment, although imagine of own movement is also possible. Kinesthetic motor imagery depends on dynamic relationship among the individual, the movement and the environment and it should be determined by the nature of the task, the environment and individual characteristics and also requires "feel" the movement.

The aim of this study is to translate this questionnaire into Turkish and the translation in terms of its internal consistency, test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* ages between 18-65 years, healthy volunteers, with no limitation in mobility or movement disorder, with no chronic pain

Exclusion Criteria:

* refuse to attend to the study, neurological conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cronbach's Alpha coefficient | 2 years
  Cronbach's Alpha coefficient was used to determine internal consistency of the questionnaire and its subscales. Cronbach's Alpha Coefficient greater than 0.8 is generally considered acceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)